CLINICAL TRIAL: NCT01028196
Title: Epidemiological Observational Non-interventional Study to Research the Prevalence of Bipolar Criteria of Hospital In-patients With Schizophrenia and Patients With Recurrent Depression
Brief Title: Observational Study to Evaluate Bipolar Disorder Symptoms in Patients Presented With Schizophrenia or Depression
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NRU-DUM-2009/1
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Recurrent Depression
Keywords: schizophrenia; schizoaffective disorder; recurrent depression; Bipolar disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Depression; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 - schizophrenia: Psychiatrists will enrol patients meeting inclusion/exclusion criteria with schizophrenia as they routinely attend the clinic or are examined in hospital in a consecutively manner.
- 2 - recurrent depression: Psychiatrists will enrol patients meeting inclusion/exclusion criteria with recurrent depression as they routinely attend the clinic or are examined in hospital in a consecutively manner.

SUMMARY:
This study is aimed to evaluate the bipolar disorder symptoms in patients presented with schizophrenia, schizoaffective disorder or recurrent depression.

Bipolar disorder is a group of mood disorders characterised by elevated or irritable mood episodes in patient's lifetime history accompanied by some additional symptoms. In this study modern bipolar disorders screening/assessment instruments will be used to explore the prevalence of bipolarity symptoms in patients who never been diagnosed with bipolar disorders. The results of this study could be useful for more accurate assessment of bipolar disorders prevalence in psychiatric patient population, could help to improve the diagnostics of bipolar disorders and management of bipolar patients.

ELIGIBILITY:
Inclusion Criteria:

* signed patient informed consent
* In-patients with the diagnosis of schizophrenia with episodic course or schizoaffective disorder, OR in-patients and out-patients with the diagnosis of recurrent depression.
* The duration of the disease is 3 years and longer and two or more episodes of the disease in the patients history.

Exclusion Criteria:

* Current diagnosis of Bipolar Disorder
* Severe and unspecified forms of schizophrenia (schizophrenia with continuous course, hebephrenic schizophrenia, catatonic schizophrenia, undifferentiated schizophrenia, unspecified schizophrenia) and organic affective disorder or intoxication induced affective disorder.
* Any other concomitant conditions which, in the judgment of investigator, will not allow the patient to complete the study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having current diagnosis of schizophrenia/ schizoaffective disorder (in-patients) and patients having current diagnosis of recurrent depression (both in-patients and out-patients) will be included into this study.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey N. Mosolov, Prof., Principal Investigator — Mental Disorders Moscow Research Institute of Psychiatry
Locations (3):
- Russia (3):
  - Research Site, Chita
  - Research Site, Moscow
  - Research Site, Novosibirsk